CLINICAL TRIAL: NCT01523132
Title: Persistent Pain After Breast Cancer Treatment (PPBCT) - Risk Factors and Pathophysiological Mechanisms
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Breast Cancer Cooperative Group (Other); Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Kenneth Geving Andersen, Physician, research fellow, Rigshospitalet, Denmark
Other Study IDs: H-D-2007-0098
Record Dates: First submitted 2012-01-27; First posted 2012-02-01 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Breast Cancer; Persistent Pain; Lymphedema; Neuropathic Pain; Neuropathy
MeSH Terms: conditions — Breast Neoplasms; Lymphedema; Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Breast cancer patients: Female breast cancer patients without metastasis and locally advanced disease

SUMMARY:
The study is a prospective cohort study following breast cancer patients from before surgery to one year after. The aims of the study are to determine risk factors that predispose to the development of persistent pain.

DETAILED DESCRIPTION:
The aim of the study is 1) to determine pre-, intra and post surgical risk factors for persistent pain after breast cancer treatment 2) to examine the prevalence of persistent pain 6 and 12 months after surgery 3) provide a quantitative sensory testing (QST) profile of the patient population, measured pre surgery, 1 week and 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with breast cancer
* 18 years or older

Exclusion Criteria:

* unable to give written consent
* unable to understand Danish
* Previous cosmetic surgery in the breast
* Previous surgery in ipsilateral breast
* Bilateral cancer
* Concomitant corrective surgery on contralateral side
* Pregnant
* Other disease or injury in the nervous system
* Psychiatric disease
* Alcohol or drug abuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients treated in a university hospital
Sampling Method: Probability Sample
Enrollment: 545 (Actual)
Dates: Start 2011-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Risk factors predisposing for persistent pain after breast cancer treatment | 12 months postoperative
  Pre-, intra- and postoperative risk factors predisposing for persistent pain

SECONDARY OUTCOMES:
Prevalence of persistent pain after breast cancer treatment | 12 months postoperative
Prevalence of sensory disturbances after breast cancer treatment | 12 months
Correlation of persistent pain after breast cancer treatment and damage of the intercostobrachial nerve | 12 months
Quantitative sensory testing: profile and correlation to persistent pain, sensory disturbances, signs of neuropathic pain, and treatment related factors | 12 months
Genetic markers and the development of persistent pain after breast cancer treatment | 12 months postoperative
QST profile 1 week after surgery for breast cancer | 1 week postoperative
  Detailed QST profile 1 week after surgery for breast cancer. Patients will be assessed with sensory mapping, followed by assessment of mechanical and thermal thresholds.
Acute pain after surgery for breast cancer | 1 week postoperative
  Prevalence of acute pain 1 week after surgery for breast cancer.
Test-Retest of QST after breast cancer treatment | 12 months postoperative
  A test-retest series of a subgroup of patients assessed with QST, to evaluate methodological reliability. Patients are scheduled to 2 QST assessments with a week between.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Geving Andersen, MD, Principal Investigator — Rigshospitalet, Denmark; Henrik Kehlet, MD, PhD, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen University Hospital, Copenhagen, Denmark

REFERENCES:
- [Background] Andersen KG, Kehlet H. Persistent pain after breast cancer treatment: a critical review of risk factors and strategies for prevention. J Pain. 2011 Jul;12(7):725-46. doi: 10.1016/j.jpain.2010.12.005. Epub 2011 Mar 24. PMID 21435953
- [Result] Andersen KG, Duriaud HM, Jensen HE, Kroman N, Kehlet H. Predictive factors for the development of persistent pain after breast cancer surgery. Pain. 2015 Dec;156(12):2413-2422. doi: 10.1097/j.pain.0000000000000298. PMID 26176893
- [Result] Andersen KG, Kehlet H, Aasvang EK. Test-retest agreement and reliability of quantitative sensory testing 1 year after breast cancer surgery. Clin J Pain. 2015 May;31(5):393-403. doi: 10.1097/AJP.0000000000000136. PMID 25084072
- [Result] Andersen KG, Duriaud HM, Aasvang EK, Kehlet H. Association between sensory dysfunction and pain 1 week after breast cancer surgery: a psychophysical study. Acta Anaesthesiol Scand. 2016 Feb;60(2):259-69. doi: 10.1111/aas.12641. Epub 2015 Oct 8. PMID 26446738
- [Result] Andersen KG, Aasvang EK, Kroman N, Kehlet H. Intercostobrachial nerve handling and pain after axillary lymph node dissection for breast cancer. Acta Anaesthesiol Scand. 2014 Nov;58(10):1240-8. doi: 10.1111/aas.12393. PMID 25307709